CLINICAL TRIAL: NCT02391493
Title: Neural Correlates of Language Control in Bilinguals. Functional MRI and Stimulation Mapping Data in Awake Surgery. (NEUROSWITCH)
Brief Title: Neural Correlates of Language Control in Bilinguals. Functional MRI and Stimulation Mapping Data in Awake Surgery.
Acronym: NEUROSWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13 245 03; HAO 2013 (Other Grant/Funding Number: Maison des sciences de l'homme de Toulouse)
Record Dates: First submitted 2015-03-04; First posted 2015-03-18 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Bilingualism
Keywords: bilinguals; language control; executive functions; functional MRI; stimulation mapping; brain tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy early bilinguals (Experimental): healthy early bilinguals functional magnetic resonance imaging
  Interventions: Device: functional magnetic resonance imaging
- healthy late bilinguals (Experimental): healthy late bilinguals functional magnetic resonance imaging
  Interventions: Device: functional magnetic resonance imaging
- bilingual patients (Experimental): bilingual patients suffering from low-grade glioma in the language areas functional magnetic resonance imaging
  Interventions: Device: functional magnetic resonance imaging

INTERVENTIONS:
Device: functional magnetic resonance imaging — Stimuli will be presented in 3 language conditions, French, English and "switch" in which the participant alternates between English and French every trial. A block design will be used, with 7 line drawings per language condition. Four 9-minute runs will be performed, there being 2 action runs and 2 object runs. In each run, there are 6 blocks of each language condition, presented in a fixed random order. No drawings are repeated. Each stimulus is preceded either by an English or a French prompt word ("to" or "faire" for actions and, "say" or "dire" for objects) for 450 msec; stimuli are presented for 1.5 seconds and followed by a blank screen for 1 second. Language blocks are separated by a variable duration (from 8 to 10 seconds).

SUMMARY:
For bilingual and multilingual patients, brain activation and Electric Stimulation Mapping studies have shown that different languages may be localized, at least partially, in distinct microanatomical systems located within the same gross anatomical areas.

The present investigation involves both types of healthy bilinguals with carefully controlled proficiency levels, as well as bilingual patients suffering from low-grade glioma.

Functional magnetic resonance imaging data will be collected while the participants perform a picture naming task in blocked conditions for both languages (either English or French) or in switch condition (English and French). A stimulation mapping study will be conducted in the patients during awake surgery with the same tasks.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Bilingual patients with a pathology indicating an intervention in awake surgery (e.g. low-grade glioma)
* At least C1-level of the CECR in both languages
* At least 12 years of schooling (French BAC)
* Right-handed (Edinburgh test, 1971)
* Performance indicator Eastern Cooperative Oncology Group 0-2 (cf. annexe)
* Life expectation > 6 month
* Affiliated to social insurance
* Having given informed consent

Healthy volunteers:

* French-English or English-French bilinguals with at least a C1 level (CECR) in both languages
* At least 12 years of schooling (French BAC)
* Right-handed (Edinburgh test, 1971)
* Early bilinguals: age of acquisition of both languages < 3 years
* Late bilinguals: age of acquisition of the L2 > 10 years

Exclusion Criteria:

Patients:

* Contra-indication for MRI
* Left-handed or ambidexter (less than +80 at the Edinburgh test - 1971)
* Mini-Mental State Examination <26
* Patient who cannot respect the procedures, visits, exams described in the protocol
* Any other medical or psychiatric affection which renders inclusion of the patient to the study inappropriate as judged by the principal investigator

Healthy volunteers:

* Contra-indication for MRI
* Mini-Mental State Examination < 26
* Age of acquisition of one of the language between 3 and 10 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Brain activity | 24 hours
  The primary judgment criteria is brain activity as measured by functional magnetic resonance imaging :
  * In blocked vs. switched naming in control subjects
  * In switched naming in early vs. late bilingual subjects
  * In blocked vs. switched naming in early vs. late bilingual subjects

SECONDARY OUTCOMES:
Brain activity | 24 hours
  The secondary judgment criteria is brain activity measured by functional magnetic resonance imaging :
  * In blocked vs. switched naming in the patients
  * In French vs. English and English vs. French naming in the late bilinguals
  * In French vs. English and English vs. French naming in the early bilinguals
  * In French vs. LX and LX vs. French naming in the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LUBRANO, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France